CLINICAL TRIAL: NCT04779333
Title: Lifestyle Enhancement for ADHD Program (LEAP) Study 2
Brief Title: Lifestyle Enhancement for ADHD Program 2
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Pooja Tandon, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002356; R33AT010041 (NIH)
Record Dates: First submitted 2021-02-24; First posted 2021-03-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEAP Group (Experimental): In addition to the components of the BMT group, the LEAP program includes an emphasis on supporting optimal physical activity, limiting screen time, and encouraging adequate sleep. The child and caregiver are also given a wrist-worn activity tracker and caregivers participate in a motivational Facebook group.
  Interventions: Behavioral: LEAP
- BMT Group (Active Comparator): The BMT Group will take part in a family-based intervention within the context of evidence-based behavioral management training (BMT) for caregivers. Standard BMT represents the current standard of care for childhood ADHD.
  Interventions: Behavioral: Standard BMT

INTERVENTIONS:
Behavioral: LEAP — LEAP will be delivered through the typical 9 weekly BMT group sessions lasting 90 minutes. Plus wrist worn activity tracker & facebook group.
  Arms: LEAP Group
Behavioral: Standard BMT — Weekly BMT groups sessions which follow the Barkley curriculum
  Arms: BMT Group

SUMMARY:
The purpose of this study is to increase physical activity (PA) in children with ADHD using a novel, family-based intervention that promotes PA within the context of evidence-based behavioral management training (BMT) for caregivers, enhanced with mobile health (mHealth) behavior change strategies.

Primary Objective: To evaluate the primary effects of a 9-week, family-based intervention (Lifestyle Enhancement for ADHD Program - LEAP) to promote PA in young children with ADHD

Secondary: To evaluate secondary effects of the LEAP program on child ADHD symptoms and executive functioning

DETAILED DESCRIPTION:
This is a randomized trial comparing the LEAP program to standard BMT for ADHD (without the enhanced focus on health behaviors, mHealth technology, or social media). Specifically, 80 families will be randomized to receive either LEAP or a standard BMT program based on Russell Barkley's Defiant Children intervention manual. Moderators (e.g., child sex, medication, BMI) and mediators (e.g., change in PA) will be analyzed as exploratory outcomes. Hypotheses being tested include: 1) LEAP will be successful in increasing PA in children with ADHD in the short-term and over a year, more so than standard BPT and 2) children randomized to LEAP will exhibit greater and more sustained improvement in clinical outcomes relative to standard BMT. If successful, the R33 phase will inform the development of a larger and longer, confirmatory trial.

ELIGIBILITY:
Inclusion Criteria (child):

* Age 6-10 years
* ADHD diagnosis
* CGI-S rating ranging from 4 to 7.
* Child not wearing a wrist-worn activity tracker more than 50% of days in the past month

Inclusion Criteria (caregiver):

* One adult custodial caregiver (resides with the child at least 50% of the time) willing to participate in the study and complete baseline/follow-up measures
* Caregiver able to complete forms in English
* Caregiver owns a smart phone or similar Garmin compatible mobile device (e.g. iPod Touch) or willing to borrow iPod from study coordinators during the study period
* Agree to install and share data from the Garmin smart phone app with investigators

Inclusion Criteria (supplementary caregiver):

* An additional caregiver designated by the participating caregiver who provides care for the participating child on at least one occasion every other week
* Able to participate in one or more group sessions
* Able to consent in English

Exclusion Criteria (children):

* - Younger than 6 years old or older than 10 years old
* Do not meet criteria currently for ADHD diagnosis
* Meet diagnostic criteria for psychiatric co-morbidities of Autism Spectrum Disorder, Depressive Disorder, Mood Disorder, Psychotic Disorder, or Intellectual Disability (by history)
* Per caregiver report, engage in >60 min/day of MVPA consistently for at least 5 days per week
* Any physical or medical restrictions on PA
* Child currently/previously used a wearable physical activity sensing device at least 50% of days in the past month

Exclusion Criteria (caregiver):

- Caregiver participated in an evidence-based parent behavior management training program (i.e., Incredible Years, Triple P, PCIT, Barkley's Defiant Child) in the past 24 months.

Exclusion Criteria (supplementary caregiver): none

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Effects of intervention on Physical Activity | Baseline to 10 weeks
  Comparing within-subject pre to post activity (MVPA) using accelerometer data
Effects of intervention on Physical Activity | Baseline to 20 weeks
  Comparing within-subject pre to post activity (MVPA) using accelerometer data
Effects of intervention on Physical Activity | Baseline to 1 year
  Comparing within-subject pre to post activity (MVPA) using accelerometer data

SECONDARY OUTCOMES:
Effects of LEAP participation on child executive function | Baseline to 10 weeks
  Evaluate effects of LEAP participation on the child's executive functioning using the parent reported BRIEF-2 measure
Effects of LEAP participation on child executive function | Baseline to 20 weeks
  Evaluate effects of LEAP participation on the child's executive functioning using the parent reported BRIEF-2 measure
Effects of LEAP participation on child executive function | Baseline to 1 year
  Evaluate effects of LEAP participation on the child's executive functioning using the parent reported BRIEF-2 measure
Effects of LEAP participation on child ADHD symptoms | Baseline to 10 weeks
  Evaluate effects of LEAP participation on the child's ADHD symptoms using the Conners-3 Parent Rating Scale
Effects of LEAP participation on child ADHD symptoms | Baseline to 20 weeks
  Evaluate effects of LEAP participation on the child's ADHD symptoms using the Conners-3 Parent Rating Scale
Effects of LEAP participation on child ADHD symptoms | Baseline to 1 year
  Evaluate effects of LEAP participation on the child's ADHD symptoms using the Conners-3 Parent Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Tandon, MD, Principal Investigator — Seattle Children's Hospital; Erin Gonzalez, PHD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States